CLINICAL TRIAL: NCT05838625
Title: A Randomized, Multicenter, 16-week Study to Evaluate the Efficacy and Safety of Two Prescription Digital Therapeutics as an Adjunct to Standard-of-Care Antipsychotic Therapy in Adult and Late Adolescent Participants With Experiential Negative Symptoms of Schizophrenia
Brief Title: Study of Two Digital Therapeutics for the Treatment of Experiential Negative Symptoms of Schizophrenia
Acronym: CONVOKE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-155-R-001
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia
Keywords: Prescription digital therapeutic (PDT); Software as a Medical Device (SaMD); Smartphone app; Schizophrenia; Negative Symptoms
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Digital Therapeutic A (Experimental): Evaluate the efficacy and safety of digital therapeutic A as an adjunct treatment to SOC in participants with experiential negative symptoms of schizophrenia.
  Interventions: Device: Digital Therapeutic
- Digital Therapeutic B (Experimental): Evaluate the efficacy and safety of digital therapeutic B as an adjunct treatment to SOC in participants with experiential negative symptoms of schizophrenia.
  Interventions: Device: Digital Therapeutic

INTERVENTIONS:
Device: Digital Therapeutic — A prescription digital therapeutic in the form of a smartphone app.

SUMMARY:
This study evaluates the efficacy of two prescription digital therapeutics (PDT) in addition to standard of care (SOC) therapy for the treatment of experiential negative symptoms of schizophrenia in late adolescents and adults.

DETAILED DESCRIPTION:
The purpose of the proposed study is to evaluate the efficacy and safety of two prescription digital therapeutics as an adjunct treatment to SOC in participants 18 years of age or older diagnosed with experiential negative symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

A participant will be eligible for entry into the study if all of the following criteria are met:

1. Has a primary diagnosis of schizophrenia.
2. Is on a stable dose of antipsychotic medication(s).
3. Has obtained an average score of ≥2 (moderate to severe) in at least two of the three CAINS-MAP domains (Social, Work, or Recreational).

Exclusion Criteria:

A participant will not be eligible for study entry if any of the following criteria are met:

1. Is currently treated with more than two antipsychotic medications (including more than two dosage forms).
2. Meets DSM-5, for diagnoses not under investigation.
3. Has participated in a CT-155 clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Experiential negative symptoms | Baseline to Week 16
  Change from baseline to Week 16 in experiential negative symptoms, as assessed by Clinical Assessment Interview for Negative Symptoms, Motivation and Pleasure Scale (CAINS-MAP)

SECONDARY OUTCOMES:
Motivation and pleasure symptoms | Baseline to Week 8
  Change from baseline in motivation and pleasure symptoms at Week 8, as assessed by CAINS-MAP
Expressive negative symptoms | Baseline to Weeks 8 and 16
  Change from baseline in expressive negative symptoms at Weeks 8 and 16, as assessed by the Clinical Assessment Interview for Negative Symptoms, Expressivity Scale (CAINS-EXP)
Positive symptoms | Baseline to Weeks 8 and 16
  Change from baseline in positive symptoms at Weeks 8 and 16, as assessed by the Positive and Negative Syndrome Scale (PANSS)
Social functioning | Baseline to Weeks 8 and 16
  Change from baseline in social functioning at Weeks 8 and 16, as assessed by the Personal and Social Performance Scale (PSP)
Self-reported defeatist beliefs | Baseline to Weeks 8 and 16
  Change from baseline in self-reported defeatist beliefs at Weeks 8 and 16, as assessed by the Defeatist Beliefs Subscale of the Dysfunctional Attitudes Scale (DAS)
Patient global impression of improvement | Weeks 8 and 16
  Patient Global Impression of Improvement Scale (PGI-I) at Weeks 8 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Viveca Livezey, MD, Study Director — Click Therapeutics
Locations (54):
- United States (54):
  - Investigational center, Chandler, Arizona
  - Investigational center, Phoenix, Arizona
  - Investigational center, Anaheim, California
  - Investigational center, Culver City, California
  - Investigational center, Garden Grove, California
  - Investigational center, La Habra, California
  - Investigational center, Long Beach, California
  - Investigational center, Los Angeles, California
  - Investigational center, Newport Beach, California
  - Investigational center, Oceanside, California
  - Investigational center, Orange, California
  - Investigational center, San Bernardino, California
  - Investigational center, Torrance, California
  - Investigational center, Cromwell, Connecticut
  - Investigational center, Hartford, Connecticut
  - Investigational center, Hialeah, Florida
  - Investigational center, Largo, Florida
  - Investigational center, Miami, Florida
  - Investigational center, Miami Lakes, Florida
  - Investigational center, Orlando, Florida
  - Investigational center, West Palm Beach, Florida
  - Investigational center, Atlanta, Georgia
  - Investigational center, Augusta, Georgia
  - Investigational center, Chicago, Illinois
  - Investigational center, Springfield, Illinois
  - Investigational center, Warrenville, Illinois
  - Investigational center, Marrero, Louisiana
  - Investigational center, Baltimore, Maryland
  - Investigational center, Boston, Massachusetts
  - Investigational center, Flowood, Mississippi
  - Investigational center, St Louis, Missouri
  - Investigational center, Omaha, Nebraska
  - Investigational center, Las Vegas, Nevada
  - Investigational center, Marlton, New Jersey
  - Investigational center, Cedarhurst, New York
  - Investigational center, Glen Oaks, New York
  - Click Therapeutics, New York, New York
  - Investigational center, New York, New York
  - Investigational center, Rochester, New York
  - Investigational center, Charlotte, North Carolina
  - Investigational center, Beachwood, Ohio
  - Investigational center, Cincinnati, Ohio
  - Investigational center, Columbus, Ohio
  - Investigational center, Oklahoma City, Oklahoma
  - Investigational center, State College, Pennsylvania
  - Investigational center, Charleston, South Carolina
  - Investigational center, Austin, Texas
  - Investigational center, Forth Worth, Texas
  - Investigational center, Houston, Texas
  - Investigational center, Irving, Texas
  - Investigational center, Mesquite, Texas
  - Investigational center, Plano, Texas
  - Investigational center, Salt Lake City, Utah
  - Investigational center, St. George, Utah

REFERENCES:
- [Derived] Lakhan SE, Dorner-Ciossek C, Besedina O, Dickerson F, Hastedt C, Isla R, Kahn RS, Lindenmayer JP, Mehta R, Snipes C, Speier A, Tang W, Willis B, Fernandez JW, von der Goltz C, Pratap A. Effectiveness, Engagement, and Safety of a Digital Therapeutic (CT-155/BI 3972080) for Treating Negative Symptoms in People With Schizophrenia: Protocol for the Phase 3 CONVOKE Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 7;14:e81293. doi: 10.2196/81293. PMID 41057039